CLINICAL TRIAL: NCT03092128
Title: Retrospective Study Based on Pharmacokinetics, Somatic Mutations and Genetic Polymorphisms Related to Individual Variations of Drug Effect and Adverse Drug Reaction of Imatinib in Gastrointestinal Stromal Tumor Treatment.
Brief Title: A Retrospective Pharmacokinetics and Pharmacogenomics Research of Imatinib in Gastrointestinal Stromal Tumor Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xueding Wang (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Xueding Wang, Institute of Clinical Pharmacology, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: SYSUCC20141021007
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Gastrointestinal Stromal Tumors; Germline Mutation; Somatic Mutation; Plasma Concentration
Keywords: Gastrointestinal stromal tumor (GIST); Imatinib; Pharmacogenetics; Pharmacokinetics; Precision medicine; Somatic and germ-line mutations
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. FFPE samples of tissue needle biopsy were used for KIT and PDGFRA mutation detection.
  2. EDTA-whole blood was centrifuged at 4000rpm*10min,plasma was separated within four hours for somatic mutation detection.The remaining samples were used for germline mutation detection. All the blood samples were frozen in -80℃ until analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sensitive group; non-sensitive group: sensitive patients were defined as patients reached CR or PR after first month administration,SD after first three months administration. non-sensitive patients were defined as patients reached PD after first month administration and first three months administration.

SUMMARY:
For patients of GIST (Gastrointestinal Stromal Tumor), Imatinib has been widely used in GIST with KIT or PDGFRA sensitive mutations. From clinical points of view, individual differences often occur between different patients, leading diverse effect in ADR and drug effect. Meanwhile, the drug effect and adverse drug reaction was significantly influenced by the pharmacokinetic factors and pharmacodynamic and other factors. In this research, we try to establish a more sensitive method to detect sensitive mutations in plasma and discover the correlation between somatic and germline mutations, plasma trough concentration and drug effect, the association between ADME-associated SNP, Target/Receptor/Pathway-associated SNP, trough concentration and TKI adverse effect. Furthermore, in vivo and in vitro research is also crucial for rational explanation for these clinical phenomenon.

DETAILED DESCRIPTION:
The plasma concentration of Imatinib were established. The ADME-associated SNPs included are CYP3A4, CYP3A4, CYP1A1, CYP2C9, CYP2C19, ABCB1, ABCG2, ABCC4, SLC22A1, SLCO1B3 and so on. The Target/Receptor/Pathway-associated SNP s included KIT, PDGFRA, PDGFRB, FLT1, FLT3, MAPK1, SHC1, CCL5, CXCL14 and so on. The somatic mutations included are KIT, PDGFRA, BRAF and so on.

ELIGIBILITY:
Inclusion Criteria:

* The main patient entry criteria included: age≥ 18 years; histologically and cytologically proved GIST; Eastern cooperative oncology group performance status (ECOGPS)≤2; adequate hematological,renal,and hepatic functions.

Exclusion Criteria:

* uncontrolled systemic disease,and other chemotherapy at the time of inclusion. The protocol was approved by the Ethical Committee of Cancer Center of Sun Yat-Sen University (CCSU), and written informed consent was obtained form each patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GIST (Gastrointestinal stromal tumor) patients; administrated with Imatinib and Sunitinib.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | The time from the date of randomisation (baseline) to the date of objective tumour progression，and expected average of 36 months.
  Excluding clinical deterioration without evidence of objective progression according to the Response Evaluation Criteria In Solid Tumors (RECIST), or death from any cause.

SECONDARY OUTCOMES:
Number of patients with objective response and adverse events | one month, three month, 12 month
  Objective responses (complete response plus partial response) and disease control (objective response plus stable disease≥6 weeks) were established according to RECIST.And adverse events was established according to CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Min Huang, Professor, Study Chair — Institute of Clinical Pharmacology, SunYat-senU
Locations (1):
- Institute of Clinical Pharmacology, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angelini S, Ravegnini G, Fletcher JA, Maffei F, Hrelia P. Clinical relevance of pharmacogenetics in gastrointestinal stromal tumor treatment in the era of personalized therapy. Pharmacogenomics. 2013 Jun;14(8):941-56. doi: 10.2217/pgs.13.63. PMID 23746188
- [Background] Demetri GD, Wang Y, Wehrle E, Racine A, Nikolova Z, Blanke CD, Joensuu H, von Mehren M. Imatinib plasma levels are correlated with clinical benefit in patients with unresectable/metastatic gastrointestinal stromal tumors. J Clin Oncol. 2009 Jul 1;27(19):3141-7. doi: 10.1200/JCO.2008.20.4818. Epub 2009 May 18. PMID 19451435
- [Background] Bouchet S, Poulette S, Titier K, Moore N, Lassalle R, Abouelfath A, Italiano A, Chevreau C, Bompas E, Collard O, Duffaud F, Rios M, Cupissol D, Adenis A, Ray-Coquard I, Bouche O, Le Cesne A, Bui B, Blay JY, Molimard M. Relationship between imatinib trough concentration and outcomes in the treatment of advanced gastrointestinal stromal tumours in a real-life setting. Eur J Cancer. 2016 Apr;57:31-8. doi: 10.1016/j.ejca.2015.12.029. Epub 2016 Feb 4. PMID 26851399
- [Background] Joensuu H, Hohenberger P, Corless CL. Gastrointestinal stromal tumour. Lancet. 2013 Sep 14;382(9896):973-83. doi: 10.1016/S0140-6736(13)60106-3. Epub 2013 Apr 24. PMID 23623056
- See also: Collaborative Innovation Center for Cancer Medicine Sun Yat-sen University Cancer Center — http://english.sysucc.org.cn/